CLINICAL TRIAL: NCT02605863
Title: The Effect of Androgen Deprivation Therapy With Enzalutamide on Bladder Cancer Chemoprevention
Brief Title: Enzalutamide for Bladder Cancer Chemoprevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment, sponsor withdrew support for study
Sponsor: University of Rochester (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Edward Messing, Principal Investigator, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 52539
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Bladder Cancer
Keywords: Enzalutamide; Non-Muscle Invasive Bladder Cancer; Androgen Deprivation Therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermediate Risk NMIBC (Experimental): Enzalutamide 160mg by mouth daily for 12 months
  Interventions: Drug: Enzalutamide
- High Risk NMIBC (Experimental): Enzalutamide 160mg by mouth daily for 12 months
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — 160 mg by mouth daily for 12 months
  Other Names: Xtandi

SUMMARY:
The purpose of this study is to examine the effect of androgen deprivation therapy through administration of enzalutamide on preventing bladder cancer recurrences in patients with non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
* A blood draw and an electrocardiogram (EKG). The blood draw will check levels of testosterone, dihydro-testosterone, estradiol, and Vitamin D. Pre-study blood-work will also include a complete blood count (CBC), basic metabolic panel (BMP/CHEM8) and liver function test (LFT) if any of these labs were not drawn within 1 month prior to the transurethral resection of bladder tumor (TURBT).
* Bladder tumor sample that is stored in the Department of Pathology will have additional tests run on it to confirm study eligibility and to test for certain cell markers.
* After 1 month following the original TURBT, subjects will begin therapy with enzalutamide. The study drug will be administered orally at a dose of 160mg daily for 12 months.
* Subjects will be monitored for adverse reactions or side effects from enzalutamide at scheduled office visits.
* If the bladder tumor is classified as being "intermediate risk", regularly scheduled office visits will occur at 2 months post-operatively (i.e., 1 month after starting enzalutamide), and then again at post-operative months 3, 6, 9 and 12, as is part of the usual standard of care.
* If the bladder tumor is classified as being "high risk" and the subject receives BCG therapy, then the office visits will occur on a slightly different schedule to conform to the standard of care for this type of disease. Subjects in this group typically start their intravesical BCG instillations 4-6 weeks post-operatively. Therefore, the subjects will be seen approximately 1 month following the initial TURBT, and will begin therapy with enzalutamide at that time, as described above. Subjects will be on study drug at least 7 days prior to the initiation of BCG therapy, which will occur once a week for 6 weeks. Similar to the subjects in the intermediate risk group, the subjects receiving BCG will also be seen 1 month after initiation of enzalutamide therapy to ensure there are no adverse reactions to the study drug. Following this visit, they will be seen again at the time of the post-BCG cystoscopy, which occurs 1 month after your 6th instillation. Subjects will be seen again at the 3, 6, 9 and 12-month post-BCG cystoscopy office visits, as part of routine care.
* Repeat blood work (CBC, BMP and LFTs) will be checked 1 month after starting enzalutamide (approximately 2 months post-operatively). For subjects with intermediate risk bladder cancer, these labs will be checked again at 3, 6, 9 and 12 months post-operatively (as per the regularly scheduled office visits). For the high risk patients receiving BCG therapy, these labs will be checked again at the 1, 3, 6 and 9-month post-BCG office visits (per the regularly scheduled office visits for these patients).
* An EKG will be obtained at baseline (before starting the study drug), but will also be re-checked at approximately 6 months (half-way through therapy with enzalutamide) to ensure there are no signs of worsening cardiac disease while on the study drug.
* A cystoscopy will be done every 3 months as part of the standard of care for bladder cancer follow-up. Lesions suspicious for tumor recurrence will be biopsied as per usual standard of care. If a recurrence is documented, subjects will discontinue use of enzalutamide.
* For subjects scheduled to undergo therapy with BCG, additional tests will be run on the urine samples that subjects will already be providing in the Urology office as part of the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed NMIBC who have undergone their TURBT.
2. Per the European Association of Urology (EAU) guidelines, only subjects with "Intermediate" or "High risk" bladder cancer will be enrolled21:

   For patients with "high risk" bladder cancer, only those who undergo BCG therapy following their TURBT will be eligible for enrollment.
3. Subjects who receive BCG instillations post-operatively will be eligible for enrollment.
4. Subjects whose tumors are AR(+) as well as AR(-) will be included, but we will restrict inclusion of AR(-) subjects so that they represent no more than 1/3 of the total study population, or any single cohort (ie. the intermediate or high-risk groups).
5. Subjects of child-bearing potential must agree to 2 acceptable forms of birth control.

Exclusion Criteria:

1. Subjects with "low risk" bladder cancer, as defined by the EAU guidelines21, will be ineligible for enrollment.
2. Subjects with "high risk" bladder cancer who do not undergo BCG therapy following their TURBT will be ineligible for enrollment.
3. Subjects who have "failed" BCG therapy in the past (had a recurrence of bladder cancer despite prior use of BCG) will be ineligible for enrollment.
4. Subjects who receive an immediate post-TURBT single instillation of intravesical chemotherapy will be ineligible for enrollment.
5. Subjects who receive a post-operative induction course of intravesical chemotherapy (ie. more than just a single immediate post-operative dose of intravesical chemotherapy) will be ineligible for enrollment.
6. Subjects who undergo blue-light/fluorescence cystoscopy will be ineligible for enrollment.
7. Subjects with a history of heart attack within the previous 12 months or who have unstable cardiovascular status will be ineligible for enrollment.
8. Subjects who have uncontrolled hypertension (for our purposes, defined as those having a systolic blood pressure > 160 documented on 2 occasions despite appropriate medical therapy) will similarly be ineligible.
9. Subjects with a history of venous thrombo-embolism (DVT/PE) within the past 3 years.
10. Subjects with a history of seizure disorders, or those with a history of stroke or transient ischemic attacks (TIA) within the previous 12 months will be ineligible.
11. Subjects with a history of liver disease whose hepatic enzymes, alkaline phosphatase or bilirubin are greater than twice the upper limit of normal will be ineligible.
12. Subjects with kidney disease with an estimated glomerular filtration rate (eGFR) < 30 will be ineligible.
13. Subjects with neutropenia will be ineligible.
14. Subjects with clinical hypogonadism, those on androgen replacement therapy, or those with prostate cancer or other diseases treated with various forms of hormonal therapy (not including 5-alpha reductase inhibitors) will also be ineligible for study enrollment.
15. Subjects who have undergone therapy for any malignancy within the past 5 years except for basal and squamous cell carcinomas of the skin will also be ineligible.
16. Subjects with prior histories of prostate cancer treated by definitive local therapy > 5 years ago will only be eligible if they have had no clinical or biochemical evidence of recurrent prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Messing, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intermediate Risk NMIBC | High Risk NMIBC
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: no participants were enrolled in the high risk NMIBC arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermediate Risk NMIBC | High Risk NMIBC | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Disease
Description: Bladder cystoscopy, urine cytology, and pathology report
Time Frame: 1 year
Population: There were no participants enrolled in the high risk arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk NMIBC | High Risk NMIBC
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no participants enrolled in the high risk arm.
Arm/Group | Intermediate Risk NMIBC | High Risk NMIBC
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate Risk NMIBC (N=1) | High Risk NMIBC (N=0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02605863/Prot_SAP_000.pdf